CLINICAL TRIAL: NCT05698901
Title: Biomarkers and Cardiac Imaging Diagnostic Assay for Monitoring Patients With Fabry Disease
Status: Recruiting | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Charles Jia-Yin Hou, Professor, Mackay Memorial Hospital
Other Study IDs: 22CT026be
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; Disease progression; Cardiac biomarkers; Therapy response
MeSH Terms: conditions — Fabry Disease; Disease Progression | interventions — agalsidase beta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: 1. 18 years or older
  2. Male or female with Fabry disease diagnosed
  3. Presence of any one of following abnormal criteria of either: 1) Cardio-specific Biomarker; 2) Abnormal elevated value of plasma Gb3 or Lyso-Gb3; 3) Electrocardiography (ECG); 4) Cardio-specific Image.
  4. ERT Treatment naïve Fabry patients
- Group B: 1. 18 years or older
  2. Male or female with Fabry disease diagnosed
  3. Presence of any one of following abnormal criteria of either: 1) Cardio-specific Biomarker; 2) Abnormal elevated value of plasma Gb3 or Lyso-Gb3; 3) Electrocardiography (ECG); 4) Cardio-specific Image.
  4. Agalsidase beta (ERT) exposed or treated Fabry patients
  Interventions: Drug: Agalsidase beta

INTERVENTIONS:
Drug: Agalsidase beta — The treatment is following local reimbursement criteria and judge by physician
  Groups: Group B

SUMMARY:
Fabry disease (FD) is a rare X-linked lysosomal storage disorder caused by deficient activity of the enzyme α-Gal A resulting from mutations affecting the GLA gene.

It is characterized by severe multi-systemic involvement that leads to major organ failure and premature death in affected men and in some women. The α-Gal A deficiency results in progressive accumulation of un-degraded glycosphingolipids, predominantly globotriaosylceramide (Gb3), within cell lysosomes throughout the body.1

In patients at the fourth to fifth decade, left ventricular hypertrophy occur usually, and myocardial infarction and heart failure develops disease progress. Life-threatening renal, cardiac, and cerebrovascular diseases are added in later decades.2,3

Fabry disease is treatable with enzyme replacement therapy (ERT). Early recognition of symptoms and diagnosis of patients at a potentially reversible stage of the disease is therefore important. To date, plasma Lyso-Gb3 is useful in the diagnosis of Fabry disease. All male with classical Fabry disease could be discerned by an elevated plasma Lyso-GL-3; All adult female patients have elevated plasma Lyso-GL-3 above normal range.4 Other study also indicated that higher lyso-Gb3 concentrations at first visit were associated with a higher event rate in the past. Men with classical FD have higher Lyso-GL-3 values compared with patients with non-classical FD and women along with an increased risk of developing complications, more severe cardiac and renal disease.5

According to a publication from Taiwan society of cariology (TSOC) expert consensus, several cardiac biomarkers including N terminal pro B type natriuretic peptide (NT-proBNP) and cardiac troponin I/T (cTNI/cTNT) have been proposed to be alternative surrogate markers of cardiac involvement in FD.6However, there is no study to analyze the relationship between all these biomarkers including lyso-Gb3 and FD cardiac manifestation or improvement of cardiac damage outcomes under ERT yet.

There is a high prevalence of the cardiac variant (IVS4+919G→A) (~1 in 1600 males) of FD in Taiwan as revealed by newborn screening programs7,8 and patients with idiopathic HCM.9 FD patients with cardiac variant need to fulfill at least two indicators as stated in "cardiac function assessment indicators of Fabry's disease cardiac variant type" with cardiac biopsy confirmed GL3 or lyso-Gb3 lipid accumulation to get local reimbursement for treatment. Cardiac biopsy is an invasive and relative dangerous procedure that some patients would refuse to take this procedure and could not get local reimbursement resulting in delay in treatment.

Therefore in the present study the investigators are aiming to identify candidate biomarkers to establish a scoring algorithm for evaluating Fabry disease progression status or treatment response and the investigators could stage patient who with more correlated biomarkers at baseline would have higher risk to develop sever clinical outcome and initiate early therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Male or female with Fabry disease diagnosed
* Presence of any one of following abnormal criteria of either: 1) Cardio-specific Biomarker; 2) Abnormal elevated value of plasma Gb3 or Lyso-Gb3; 3) Electrocardiography (ECG); 4) Cardio-specific Image.
* Group A: ERT Treatment naïve Fabry patients
* Group B: Agalsidase beta (ERT) exposed or treated Fabry patients
* Willing and able to comply with the required clinic visits, study procedures and assessments

Exclusion Criteria:

* Patient who are unwilling to sign inform consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed FD patients with cardiac manifestation will be included and classified into two group based on their treatment status: treatment naïve or treated. Treatment naïve patient will be assigned to group A; Treated patient will be assigned to group B. If patient from group A meet the treatment criteria and about to have ERT, he/she could be re-assigned to group B.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
To establish a comprehensive scoring algorithm to evaluate the disease progression status and potential indicators in response to treatment outcome mainly from imaging or biomarkers. | 3 years

SECONDARY OUTCOMES:
(a)To figure out which biomarker and imaging data is statistically significant associated with disease progression status in patients without treatment. | 3 years
To further analyze and confirm from (a) that treatment outcomes (biomarkers/imaging parameters) of patient exposed to agalsidase beta therapy were statistically significant. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Jia-Yin Hou, Study Chair — Mackay Memorial Hospital
Locations (1):
- Charles Jia-Yin Hou, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided